CLINICAL TRIAL: NCT01857830
Title: The Effect of a Short Term Meditation Retreat on Markers of Cellular Stress and Aging
Brief Title: The Relaxation vs. Retreat Study
Acronym: R&R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-1039
Record Dates: First submitted 2013-04-25; First posted 2013-05-20 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Stress; Ageing; Wellbeing
Keywords: Telomerase; Telomere Length; Psychological Stress; Amyloid beta proteins; Meditation
MeSH Terms: conditions — Stress, Psychological; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meditation Retreat Group (Experimental): Participants in this group will participate in a 6 day meditation retreat at the La Costa Resort and Spa in Carlsbad, CA. They will be self-selected to participate in the retreat or are novice meditators randomized into this retreat.
  Interventions: Behavioral: Meditation Retreat
- Relaxation/Control Group (Active Comparator): Participants in this group will stay at La Costa Resort and spa for a 6 day period and will participate in the Active Comparator Relaxation Group activities (i.e. series of lectures on longevity and health, shared meals, and other leisure activities).
  Interventions: Behavioral: Active Comparator Relaxation Group

INTERVENTIONS:
Behavioral: Meditation Retreat — The intervention is a one week meditation and yoga retreat hosted at the La Costa Resort and Spa in Carlsbad, CA.
  Arms: Meditation Retreat Group
Behavioral: Active Comparator Relaxation Group — Participants are randomized to stay at La Costa Resort and Spa for 6 days. Participants will receive daily meals similar to the meals for those in the retreat group. Participants will also receive a daily one hour lecture on topics related to longevity and health.
  Arms: Relaxation/Control Group

SUMMARY:
The purpose of this research study is to examine whether a short term meditation intervention can improve health, mood, and biological markers of cellular stress and aging in novice and experienced meditators compared to controls.

DETAILED DESCRIPTION:
There are 3 parts to this research study, Part A, B, and C.

In Part A, participants complete a brief online questionnaire sent to them via email by the study coordinator.

During Part B of the study, participants stay at La Costa Resort in Carlsbad, CA for 6 nights and participate in a meditation retreat being held at the resort, or stay at the resort without participating in the retreat. During their stay, participants attend two in-person research assessments throughout the week. Assessments will be 4 days (96 hours) apart for all participants and will include a fasting blood draw, body measurements, and self-report questionnaires.

Part C of the study includes a brief online questionnaire that is completed 1 month after participants leave La Costa Resort.

This study includes 3 groups: a group of "novice meditators" from the greater San Diego Region that are randomized into either the 1) Relaxation (Control) group or 2) Retreat group. The third group is comprised of self-selected "experienced meditators" who are already enrolled in the retreat. In total, 99 participants were recruited for this study.

The Retreat group stays at La Costa Resort and attends a 6 day meditation retreat intervention as well as completes all research study assessments and questionnaires.

The Relaxation (Control) group stays at La Costa Resort for 6 nights, but does not attend the meditation retreat. They attend once daily lectures on science topics and complete all research study assessments and questionnaires.

The Experienced Retreat group participants have an ongoing meditation practice and have enrolled themselves in the April 2013 meditation retreat. All of the Experienced meditators attend the meditation retreat and complete all research study assessments and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Women
* Age 30-60
* "Novice Meditator" (meditates for 30 minutes per week or less) or "Experienced Meditator" (meditates at 40 or more per week and for more than 6 months, and are self-selected/enrolled in the retreat)

Exclusion Criteria:

* Current or history of a major medical condition (such as cancer, heart disease, autoimmune disease, diabetes)
* Smokers (have not smoked regularly for the past 6 months)
* Currently taking antidepressants
* Post Traumatic Stress Disorder
* Currently taking Hormone Replacement Therapy or birth control pills

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Telomerase | Change from Baseline in Telomerase 96 hours later
  Participants blood will be drawn by licensed phlebotomist on the day after their arrival at La Costa Resort at their baseline assessment and again 96 hours later at their follow-up assessment. Telomerase will be measured at both time points.

SECONDARY OUTCOMES:
Amyloid Beta Proteins | Change from baseline in Amyloid Beta Proteins, 96 hours later
  Participants blood will be drawn by licensed phlebotomist on the day after their arrival at La Costa Resort at their baseline assessment and again 96 hours later at their follow-up assessment. Amyloid beta protein levels will be measured in the blood at both time points.
Psychological Well being | Change from Baseline in psychological well being at 96 hours, and 1 month later.
  We will collect self reported measures of vitality, purpose in life, perceived stress, rumination, self-compassion, mindfulness, presence in the moment, mind wandering, depression, acceptance and action, and body responsiveness in questionnaires. Participants complete questionnaires before arriving at La Costa (baseline), after their stay (follow-up) and one month after they leave (1-month follow-up). Additionally, they complete daily questionnaires that ask about their daily experiences (emotions, stress).
Oxytocin | Change from baseline in Oxytocin at 96 hours later.
  Plasma is saved from baseline and 96 hour followup for oxytocin assays.
Telomere Length | Change from Baseline in Telomere Length, 96 hours later
  Participants blood will be drawn by licensed phlebotomist on the day after their arrival at La Costa Resort at their baseline assessment and again 96 hours later at their follow-up assessment. Telomere Length will be measured at both time points.
Gene Expression | Change from Baseline in Gene Expression, 96 hours later
  Participants blood will be drawn by licensed phlebotomist on the day after their arrival at La Costa Resort at their baseline assessment and again 96 hours later at their follow-up assessment. Patterns of gene expression (specifically on genes related to aging) will be measured at both time points.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco; Eli Puterman, PhD, Principal Investigator — University of California, San Francisco; Elizabeth Blackburn, PhD, Principal Investigator — University of California, San Francisco; Jue Lin, PhD, Principal Investigator — University of California, San Francisco; Samantha Schilf, BA, Study Director — University of California, San Francisco
Locations (1):
- Chopra Center for Wellbeing, Carlsbad, California, United States